CLINICAL TRIAL: NCT04076254
Title: Albumin 5% as Resuscitation in Adult Dengue Fever Patients With Plasma Leakage
Brief Title: Resuscitation With Albumin 5% in Dengue Haemorrhagic Fever
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Rika Bur, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DEN-09
Record Dates: First submitted 2016-10-31; First posted 2019-09-03 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Dengue Hemorrhagic
Keywords: albumin 5%; resuscitation
MeSH Terms: conditions — Dengue | interventions — Albumins; Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- albumin (Experimental): albumin 5%
  Interventions: Drug: Albumins
- fluid (Active Comparator): Ringer Lactate
  Interventions: Drug: Fluid

INTERVENTIONS:
Drug: Albumins — albumin 5%
  Arms: albumin
Drug: Fluid — Ringer Lactate
  Arms: fluid

SUMMARY:
Endothelial cell had important role in plasma leakage process. Plasma leakage occurs due to increased vascular permeability caused by disruption of endothelial glycocalyx showed by increased syndecan-1 level in serum. Endothelial vascular permeability disruption may cause several clinical manifestations such as increased haematocrit level, pleural effusion, ascites, hypoalbuminemia, thrombocytopenia, and bleeding manifestation. This condition will lead to hypoperfusion in the tissue and microvascular dysfunction. Microvascular dysfunction activated anaerob mechanism and resulting increased lactate level serum. Severe dysfunction can lead to shock and death if fluid resuscitation is inadequate in the first 24 hour.

Fluid administration becomes key therapy for plasma leakage. Crystalloid is an isotonic fluid which can fill intravascular, however this fluid also quickly moved toward extravascular. Albumin 5% can help reduce the extravasation because of it can increase the osmotic pressure and maintaining the intravascular volume. In the first 24 hour after albumin administration, albumin is hypothesized can restore intravascular volume, repair and maintain glycocalyx, maintain vascular permeability, and restore microcirculation perfusion. This mechanisms can prevent worse outcome and hoped can reduce hospital stay.

Many studies had been done regarding the choice of resuscitation fluid in septic patient. Until now, the role of albumin 5% as resuscitation fluid in DHF to prevent severe plasma leakage has not been studied.

DETAILED DESCRIPTION:
This study is an open label randomized control trial with concealment procedure which is to compare the effect of albumin 5% and ringer lactate towards plasma leakage incidence in adult DHF patient. This clinical trial cannot be done in double blind because it is technically impossible.

This study was conducted in dengue fever patients who were treated in internal medicine wards in RSUD Tangerang Selatan and RSAB Harapan Kita. Recruitment starts from October 2016 to February 2017.

The target population of this research is all adult dengue virus infected patients that were hospitalized in the hospital. Accessible population are all dengue fever patients who were treated in internal medicine wards in RSUD Tangerang Selatan and RSAB Harapan Kita from October 2016 to February 2017. Subject is accessible population that met the inclusion criteria.

All subjects who met the inclusion criteria were included in the study by consecutive sampling.

The subject allocation was done by a third party using randomized block by software WINPEPI, with the same number of subjects in each block. Randomization process will be stratified according to study sites (RSUD Tangerang Selatan and RSAB Harapan Kita).

Results of randomized translated into a sealed envelope that is not transparent. The number of envelopes in accordance with the prediction of the number of subjects in each flashlight. On the outside of the envelope is written flashlight and a number indicating the order of subject recruitment. Inside the envelope is written the type of fluid to be administered. This envelope will be opened by investigators with the witness when the subject had to be given fluid therapy. This procedure will be documented in the minutes of opening the envelope.

Researchers cooperate with doctors / paramedics at polyclinic and emergency room. Their jobs are to provide information to the researchers about the patients who infected with dengue virus proven by NS1 positive test result. Inclusion criteria based on the laboratory test are lactate ≥ 2.5 mmol/L, increased of haematocrit ≥ 10% but ≤ 15% from base line, and with or without pleural effusion and or ascites proven by abdominal ultrasound. After the subjects fulfill these inclusion criteria, researchers will proceed to do the follow-through assessment.

Subjects are given the explanation about the aim of the research, examination procedures, therapy, follow-up and side effects which may occur during the research and the benefit of participating. If the subject or family of subject approves to participate in the research, they will be given an approval form which is signed before the research conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 and ≤ 60 years
2. Patients with a history of fever ≤ 3 days, with NS1 positive, and diagnosed with DHF which marked by plasma leakage in microvascular that characterized by lactate levels ≥ 2.5 mmol / L and increased haematocrit ≥ 10% but ≤15 % of initial haematocrit. And may or not be accompanied by the presence of pleural effusion or ascites in abdominal ultrasound.
3. Patients are hospitalized at RSUD Tangerang Selatan, RS Hermina Ciputat, RSUD Cengkareng,RSUD Taman Sari, RSUD Kembangan, and RS Royal Taruma from January 2018 to February 2019.

Exclusion Criteria:

1. Patients who are pregnant and confirmed by tests β HCG, or in menstruation cycle.
2. Patients with comorbid diseases such as metabolic syndrome, liver cirrhosis, sepsis, renal disorders, hematological disorders, immunocompromised, and malnutrition.
3. Refuse to participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Syndecan-1 level | first 4 hour
  Level of Syndecan-1 in the first 4 hours after fluid resuscitation
Syndecan-1 level | first 12 hour
  Level of Syndecan-1 in the first 12 hours after fluid resuscitation
Syndecan-1 level | first 24 hour
  Level of Syndecan-1 in the first 24 hours after fluid resuscitation

SECONDARY OUTCOMES:
haematocrit level | first 4, 12, and 24 hour
  Hematocrit value in the first 4, 12, and 24 hours after fluid resuscitation
platelet count | first 4, 12, and 24 hour
  Platelet count in the first 4, 12, and 24 hours after fluid resuscitation
albumin level | first 24 and 48 hour
  Level of serum albumin in the first 4, 12, and 24 hours after fluid resuscitation
quantitative urinary protein level | first 24 and 48 hour
  Quantitative urinary protein level in the first 24 and 48 hours after fluid resuscitation
lactate level | first 12 and 24 hour
  Serum lactate level in the first 12 and 24 hours after fluid resuscitation
length of hospital stay | throughout study completion, an average of 5 days
  Patients' length of hospital stay through study completion

CONTACTS AND LOCATIONS:
Locations (1):
- RSAB Harapan Kita, Jakarta, Indonesia

REFERENCES:
- [Derived] Bur R, Suwarto S, Pohan HT, Prihartono J, Harahap AR, Dewi BE, Sadikin M, Rachman A, Yusuf H. Early intervention of 5% albumin shown superior control of vascular integrity and function compared to ringer's lactatein hospitalized adult with grade I & II Dengue hemorrhagic fever: a multicenter randomized controlled trial in Indonesia. Trop Dis Travel Med Vaccines. 2024 Oct 1;10(1):20. doi: 10.1186/s40794-024-00230-3. PMID 39350232